CLINICAL TRIAL: NCT05944601
Title: Exploring to Remediate Behavioral Disturbances of Spatial Cognition in Community-dwelling Senior Citizens With Mild Cognitive Impairment by Innovative Technological Apparatus.
Brief Title: Exploring to Remediate Behavioral Disturbances of Spatial Cognition
Acronym: BDSC-MCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03A203
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Spatial Navigation
Keywords: spatial navigation; Alzheimer's disease; mild cognitive impairment; subjective cognitive decline; elderly; APOE; assistive technology
MeSH Terms: conditions — Spatial Navigation; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy controls (No Intervention): Elderly people without cognitive impairment or subjective cognitive decline.
- Subjective cognitive decline (No Intervention): Individuals presenting cognitive complains that are not confirmed by neuropsychological testing.
- patients with MCI due to AD (Experimental): Patients with Mild Cognitive Impairment with abnormal spinal fluid test for amyloid beta protein.
  Interventions: Behavioral: Virtual and computer-based cognitive remediation training

INTERVENTIONS:
Behavioral: Virtual and computer-based cognitive remediation training — Amyloid-positive MCI patients, and individuals carrying the ApoE- ε4 allele will undergo a combined intervention of computer-based sessions of a spatial memory task by the Erica software (Giunti, Florence, Italy) and VR navigation sessions by the NeuroVirtual 3D software (Serino et al., 2010), in order to improve spatial memory for landmarks location and mental frame syncing for supporting spatial scenarios, respectively. The intervention will last one month for a total of 12 sessions (3 days a week, 50 minutes per session).
  Arms: patients with MCI due to AD

SUMMARY:
Spatial navigation (SN) has been reported to be one of the first cognitive domains to be affected in Alzheimer's disease (AD), which occurs as a result of progressive neuropathology involving specific brain areas. Moreover, the epsilon 4 isoform of Apolipoprotein-E (APOE-ε4) has been associated with both sporadic and familial late-onset AD and patients with Mild Cognitive Impairment (MCI) due to AD are more likely to progressively deteriorate. It will be investigated (i) whether amyloid-positive MCI patients and APOE-ε4 carriers show subtle changes of SN prior to the overt symptoms of AD disorientation, both in virtual and in naturalistic open-space tasks, and (ii) the effect of a combined treatment of computer-based and virtual reality tasks in those presenting such an impairment. Finally, (iii) threshold algorithms based on physiological parameters and gait analysis will be set up to support senior citizens at increased risk in maintaining their ability to independently navigate urban environments. Different types of navigational guidance will be examined on a sample of 76 older adults by the AppleGame, and the Detour Navigation Test-modified version. It is expected that patients with MCI due to AD and APOE-ε4 carriers show reduced SN performances than individuals with subjective cognitive impairment and healthy controls in the experimental tasks, with potential improvements after cognitive rehabilitation. Altered SN performances of individuals at increased risk to develop AD may inform future advanced technological applications in providing valuable information on threshold algorithms based on physiological parameters and gait analysis during elders' traveling to unfamiliar locations.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is characterized by a progressive deterioration of cognitive functions with episodic memory loss and spatial disorientation (SD) as main features. Getting lost in community due to AD is associated with a wide range of negative consequences, such as a strong decrease in patients' quality of life. Episodes of SD in the elderly can increase the possibility of being recovered in a nursing home, caused by a loss of the sense of autonomy as well as an increase in potential injuries and, in the worst cases, even death. Additionally, caregiver burden and increased stress, as well as scarce community resources represent other significant problems related to patients' SD. New technological solutions, such as virtual reality (VR), represent promising means for AD assessment and intervention, especially when they can reveal poor ecological performances. In addition to the advanced age, the ε4 allele of Apolipoprotein-E (APO-E) represents the most important risk factor for AD, providing the opportunity to evaluate subclinical behavioral alterations in individuals with subjective cognitive decline (SCD), and Mild Cognitive Impairment (MCI) due to AD, which represents the prodromic phase of dementia. Deterioration of spatial navigation (SN) abilities is often present early in the course of AD. Therefore, a better understanding the neural mechanisms related to SN impairment in patients at high risk of developing AD can help timely diagnosis and intervention. The present study, adopting a technological apparatus for the detection and the rehabilitation of SN deficits, aims to: (i) investigate the performances obtained on SN tasks in a sample of community-dwelling older adults grouped into three levels (healthy controls, individuals with SCD and patients with MCI due to AD), undergoing virtual (The AppeGame) and naturalistic open-space tests (Detour Navigation Test-modified version); (ii) correct SN deficits by computer-based cognitive remediation sessions and VR sessions; (iii) educate participants at high risk of developing dementia about the opportunity offered by technology in supporting SN in exploring urban circuits.

We will analyze results of the virtual and ecological tasks of SN as a function of age, ApoE genotype and belonging of one the three groups, using a multiple linear regression model. The subgroups of participants at highest risk of developing AD will be administered the aforementioned combined cognitive rehabilitation sessions, with a test/retest analysis. Finally, through an online technological monitoring system, participants will be provided personalized feedbacks via smartphone digital health applications connected to a wearable equipped with sensors, in order to self-manage during their journeys alone in urban environments thanks to the use of threshold algorithms capable of supporting their SN.

ELIGIBILITY:
Inclusion Criteria:

* age over 65 years;
* education not less than 5 years;
* basic ICT skills measured by the Catholic University devoted software

Exclusion Criteria:

* presence of visual, hearing or motor impairment significantly interfering with spatial navigation tasks;
* neurological/psychiatric disease or other medical conditions preventing spatial navigation;
* history of alcohol or drugs addiction;
* intake of psychotropic drugs;
* presence of dementia.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Detecting drop errors (DEs) and composite disorientation score (CDS) in individuals at increased risk to develop AD in virtual and naturalistic spatial navigation tasks, respectively | March-November 2023
  Lower performances in virtual navigation tasks (higher DEs) and in naturalistic navigation (CDS>1) in patients with MCI due to AD and in APOE-e4 carriers than healthy controls and individuals with subjective cognitive decline

SECONDARY OUTCOMES:
Improving spatial memory after a combined cognitive training (virtual reality and computer-based cognitive remediation) in a subgroup of patients with MCI due to AD and APOE-e4 carriers | December 2023-January 2024
  Higher performances in the Corsi learning Suvra-span test

OTHER OUTCOMES:
To educate a dyad (subject and caregiver) about the usefulness of a portable assistive technology for spatial navigation in community settings | January 2023-February 2024
  High scores in the Tele-healthcare Satisfaction Questionnaire-Wearable Technology

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Lombardy, Italy